CLINICAL TRIAL: NCT00367536
Title: An Open-label, Single-dose, Randomized-to-sequence, 4-period Crossover Bioavailability Study of Bazedoxifene Contained in Bazedoxifene/Conjugated Estrogen Tablets Administered to Healthy Postmenopausal Women.
Brief Title: Study Evaluating Three Bazedoxifene/Conjugated Estrogens Combination Tablet Formulations Versus BZA Oral Solution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: 3115A1-115
Record Dates: First submitted 2006-08-21; First posted 2006-08-23 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2009-07

CONDITIONS: Postmenopause
Keywords: Health
MeSH Terms: interventions — bazedoxifene

INTERVENTIONS:
Drug: bazedoxifene/conjugated estrogens combination tablet

SUMMARY:
This study involves the experimental drug bazedoxifene acetate/conjugated estrogens (also called BZA/CE). This drug is not approved by the Food and Drug Administration (FDA).

About 24 subjects will take part in this study. Each subject's participation in this study will last for about 10 weeks. During this study, each subject will receive 3 different types of BZA/CE tablets plus an oral solution containing only BZA. The purpose of this study is to learn how the tablet dosage forms dissolve and are absorbed by the body compared to the BZA oral solution. In addition, information will also be learned about the safety and tolerability of these dosage forms given to healthy postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy, nonsmoking (or smoker of less than 10 cigarettes/day)
* Postmenopausal women aged 35 to 70 years
* At least 12 months of spontaneous amenorrhea, OR 6 months of spontaneous amenorrhea with follicle-stimulating hormone (FSH) levels at least 38 mIU/mL
* Women 55 years of older must have at least 12 months of amenorrhea
* Body mass index in the range of 18.0 to 35.0, with a minimum body weight of 50 kg

Exclusion Criteria:

* A history or active presence of clinically important medical disease.
* History or alcoholism or drug abuse within 1 year before study start.
* Use of estrogen-, androgen-, or progestin-containing medication by a non-oral route of administration within 6 months before study day 1 must be approved by Wyeth Research

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2006-08; Study Completion 2006-08

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer